CLINICAL TRIAL: NCT00616343
Title: Pilot Study of Zonisamide in the Treatment of Essential Tremor
Brief Title: Zonisamide in the Treatment of Essential Tremor
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Principal Investigator left the study site on December 28, 2012.
Sponsor: Loma Linda University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: OSR#53157
Record Dates: First submitted 2008-02-04; First posted 2008-02-15 (Estimated); Results first posted 2014-07-17 (Estimated); Last update posted 2014-07-17 (Estimated); Status verified 2014-07

CONDITIONS: Essential Tremor
Keywords: ET
MeSH Terms: conditions — Essential Tremor | interventions — Zonisamide

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Zonisamide (Active Comparator)
  Interventions: Drug: Zonisamide

INTERVENTIONS:
Drug: Zonisamide — 100mg tablets once a day for two weeks, then increased to 200mg qhs for two weeks.
  Other Names: Zonegran

SUMMARY:
The purpose of this study is to determine if Zonisamide is effective in reducing tremors in patients with Essential Tremor.

DETAILED DESCRIPTION:
The subjects will remain on their usual medication and a baseline assessment using the Fahn Tolosa Marin tremor rating scale will be performed and will be video taped.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Essential Tremor based on the Tremor Investigational Group criteria for definite or probable Essential Tremor.
2. Age: 18 years or over.
3. Willingness and ability to comply with the study requirements and give informed consent.

Exclusion Criteria:

1. Known history of psychiatric disorder, major depression, dementia, aplastic anemia, or Stevens-Johnson syndrome.
2. Known alcohol or substance abuse in previous 12 months.
3. Positive pregnancy test.
4. Unwillingness to use adequate contraceptive methods if of childbearing potential.
5. Known allergy to sulfonamides.
6. Laboratory abnormalities prior to onset of trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2003-06; Primary Completion 2012-10 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David M Swope, MD, Principal Investigator — Loma Linda University

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Zonisamide
Started | 9
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: •<=18 years Male/Female Hx essential tremor
Arm/Group | Zonisamide
Number analyzed (Participants) | 9
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.1 (16.33078)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Tremor Severity
Description: PI has left the institution and we are unable to accurately assess the data from the remaining records.
Time Frame: 4 weeks
Arm/Group | Zonisamide
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Zonisamide
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 0/9

LIMITATIONS AND CAVEATS:
PI has left the institution and we are unable to accurately assess the data from the remaining records.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes